CLINICAL TRIAL: NCT06079294
Title: Impact of Confirmed Autoimmune Encephalitis on Brain Glucose Metabolism : a Prospective FDG PET Study
Brief Title: Impact of Confirmed Autoimmune Encephalitis on Brain Glucose Metabolism
Acronym: ENCEPHATAIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: APHP221163
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Autoimmune Encephalitis
Keywords: Autoimmune Encephalitis; PET; FDG; NMDAr; LGI1; CASPR2; GAD
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System; Cortical Dysplasia-Focal Epilepsy Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FDG PET (Experimental)
  Interventions: Other: FDG PET

INTERVENTIONS:
Other: FDG PET — Brain FDG PET performed 3 months after treatment initiation

SUMMARY:
Prospective cohort study evaluating FDG PET in 56 patients with confirmed autoimmune encephalitis - based on 2016 Graus criteria, and 2021 paraneoplastic neurological syndromes criteria - at the acute phase, before immunomodulating treatment, or within 10 days of treatment initiation.

DETAILED DESCRIPTION:
Autoimmune encephalitis is a diagnostic challenge, and requires early diagnosis for improved neurological outcomes. FDG PET has shown very high sensitivity, suggesting better performances than MRI, but almost exclusively in small sized retrospective studies. Brain FDG PET is therefore not included in current diagnostic criteria, conversely to brain MRI. This study will include 56 patients with confirmed - seropositive or seronegative - autoimmune encephalitis, based on 2016 Graus criteria for autoimmune encephalitis and 2021 criteria for paraneoplastic neurological syndromes. The main objective is to conduct a prospective evaluation of the diagnostic value of FDG PET performed in the acute phase before treatment initiation, or within 10 days of treatment initiation. A follow-up PET performed 3 months after treatment initiation will also be performed and analysed for all patients as part of secondary objective analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Newly diagnosed autoimmune encephalitis based on at least 1 of the 3 following criteria :

  1. " Definite limbic autoimmune encephalitis " according to 2016 Graus et al. criteria
  2. " Possible autoimmune encephalitis " according to 2016 Graus et al. criteria AND typical autoantibody detected in serum or CSF
  3. " Probable or certain paraneoplastic neurological syndrome " according to Graus et al. 2021 criteria (excluding peripheral neurological syndromes)
* Less than 6 months since first neurological symptoms imputable to autoimmune encephalitis
* Affiliated or entitled to a social security system (except AME)
* Obtaining free, written and informed consent (patient or legal representative or the close relative)

Exclusion criteria

* History of brain tumor, head trauma, infarction or cerebral hematoma likely to result in altered cerebral carbohydrate metabolism on PET
* Patients who hae been on immunotherapy (corticosteroid bolus, IVIg, plasma exchange, endoxan, rituximab or other immunotherapy) fr more than 10 days
* Pregnant or breast-feeding woman
* Ventilated intubated patient
* Absolute contraindication to MRI (Pacemaker, cochlear implant, etc.)
* Presence of cognitive disorders incompatible with goog cooperation with the PET scan
* Algic or agitated patient unable to remain immobile in supine position for 30 minutes
* Deprived of liberty or under a protective measure (guardianship or curatorship)
* Patient taking part in other interventional research involving radiopharmaceutical injections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Main analysis of initial brain FDG PET | PET performed at the acute phase, before immunomodulating treatment (or within 10 days of treatment initiation)
  Automated region-based and voxel wise quantitative PET analysis, estimation of the proportion of patients with PET anomalies (overall and by region of interest).

SECONDARY OUTCOMES:
Analysis of follow-up brain FDG PET | PET performed 3 months after treatment initiation, compared to initial brain PET
  Automated region-based and voxel wise quantitative PET analysis comparatively to initial brain PET
Secondary analysis of initial brain FDG PET | PET performed at the acute phase, before immunomodulating treatment (or within 10 days of treatment initiation)
  Subgroup PET analysis according to autoantibody subtype or seronegative status
Secondary analysis of initial brain FDG PET | PET performed at the acute phase, before immunomodulating treatment (or within 10 days of treatment initiation)
  Correlation of main analysis results to important clinical variables (clinical symptomatology (typology and duration of symptoms), MRI, cerebrospinal fluid (CSF), electroencephalogram (EEG).)
Secondary analysis of initial brain FDG PET | PET performed at the acute phase, before immunomodulating treatment (or within 10 days of treatment initiation)
  PET voxel-wise connectivity analysis
Secondary analysis of initial and follow-up brain FDG PET | PET performed at the acute phase, before immunomodulating treatment (or within 10 days of treatment initiation), and follow-up PET 3 months after treatment initiation
  Correlation of PET treatment response to clinical symptom treatment response
Analysis of initial whole body FDG PET | PET performed at the acute phase, before immunomodulating treatment (or within 10 days of treatment initiation)
  Evaluation of whole body FDG PET diagnostic performance for identifying neoplasms in paraneoplastic syndromes

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie Kas, Pr, Principal Investigator — Hôpital Pitié Salpêtrière - Assistance Publique Hôpitaux de Paris
Locations (1):
- Hospital Pitie Salpetriere, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients. Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.